CLINICAL TRIAL: NCT04451772
Title: A Phase 2, Long-Term Extension (LTE) Study With Elsubrutinib and Upadacitinib Given Alone or in Combination (ABBV-599) in Subjects With Moderately to Severely Active Systemic Lupus Erythematosus Who Have Completed the M19-130 Phase 2 Randomized Controlled Trial (RCT)
Brief Title: A Study of the Safety of Oral Elsubrutinib Capsules and Oral Upadacitinib Tablets Given Alone or in Combination (ABBV-599) for Adult Participants With Moderately to Severely Active Systemic Lupus Erythematosus to Assess Change in Disease State
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M20-186; 2020-001690-72 (EudraCT Number)
Record Dates: First submitted 2020-06-29; First posted 2020-06-30 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Systemic Lupus Erythematosus; ABBV-599; ABBV-105; ABT-494; Elsubrutinib; Upadacitinib
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) -> ABBV-599 High Dose (Experimental): Participants received elsubrutinib 60 mg capsules once a day by mouth and upadacitinib 30 mg film-coated tablets once a day by mouth for 48 weeks in Study M19-130. Participants continued on this regimen in the current study (M20-186) for up to 56 weeks.
  Interventions: Drug: Elsubrutinib; Drug: Upadacitinib
- Elsubrutinib placebo/upadacitinib 30 mg -> Elsubrutinib placebo/upadacitinib 30 mg (Experimental): Participants received placebo capsules for elsubrutinib once a day by mouth and upadacitinib 30 mg film-coated tablets once a day by mouth for 48 weeks in Study M19-130. Participants continued on this regimen in the current study (M20-186) for up to 56 weeks.
  Interventions: Drug: Placebo for Elsubrutinib; Drug: Upadacitinib
- Elsubrutinib placebo/upadacitinib placebo -> ABBV-599 High Dose (Experimental): Participants received placebo capsules for elsubrutinib once a day by mouth and placebo film-coated tablets for upadacitinib once a day by mouth for 48 weeks in Study M19-130. Participants received elsubrutinib 60 mg capsules once a day by mouth and upadacitinib 30 mg film-coated tablets once a day in the current study (M20-186) for up to 56 weeks.
  Interventions: Drug: Elsubrutinib; Drug: Upadacitinib
- ABBV-599 Low Dose (Elsubrutinib 60 mg/upadacitinib 15 mg) -> ABBV-599 Low Dose (Experimental): Participants received elsubrutinib 60 mg capsules once a day by mouth and upadacitinib 15 mg film-coated tablets once a day by mouth for 48 weeks in Study M19-130. Participants continued on this regimen in the current study (M20-186) for up to 56 weeks.
  Interventions: Drug: Elsubrutinib; Drug: Upadacitinib
- Elsubrutinib 60 mg/upadacitinib placebo -> Elsubrutinib 60 mg/upadacitinib placebo (Experimental): Participants received elsubrutinib 60 mg capsules once a day by mouth and placebo film-coated tablets for upadacitinib once a day by mouth for 48 weeks in Study M19-130. Participants continued on this regimen in the current study (M20-186) for up to 56 weeks.
  Interventions: Drug: Elsubrutinib; Drug: Placebo for Upadacitinib
- Elsubrutinib placebo/upadacitinib placebo -> ABBV-599 Low Dose (Experimental): Participants received placebo capsules for elsubrutinib once a day by mouth and placebo film-coated tablets for upadacitinib once a day by mouth for 48 weeks in Study M19-130. Participants received elsubrutinib 60 mg capsules once a day by mouth and upadacitinib 15 mg film-coated tablets once a day by mouth for 48 weeks in the current study (M20-186) for up to 56 weeks.
  Interventions: Drug: Elsubrutinib; Drug: Upadacitinib

INTERVENTIONS:
Drug: Elsubrutinib — Capsule; Oral
  Other Names: ABBV-105
  Arms: ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) -> ABBV-599 High Dose; ABBV-599 Low Dose (Elsubrutinib 60 mg/upadacitinib 15 mg) -> ABBV-599 Low Dose; Elsubrutinib 60 mg/upadacitinib placebo -> Elsubrutinib 60 mg/upadacitinib placebo; Elsubrutinib placebo/upadacitinib placebo -> ABBV-599 High Dose; Elsubrutinib placebo/upadacitinib placebo -> ABBV-599 Low Dose
Drug: Placebo for Elsubrutinib — Capsule; Oral
  Arms: Elsubrutinib placebo/upadacitinib 30 mg -> Elsubrutinib placebo/upadacitinib 30 mg
Drug: Upadacitinib — Film-coated tablet; Oral
  Other Names: ABT-494; RINVOQ
  Arms: ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) -> ABBV-599 High Dose; ABBV-599 Low Dose (Elsubrutinib 60 mg/upadacitinib 15 mg) -> ABBV-599 Low Dose; Elsubrutinib placebo/upadacitinib 30 mg -> Elsubrutinib placebo/upadacitinib 30 mg; Elsubrutinib placebo/upadacitinib placebo -> ABBV-599 High Dose; Elsubrutinib placebo/upadacitinib placebo -> ABBV-599 Low Dose
Drug: Placebo for Upadacitinib — Film-coated tablet; Oral
  Arms: Elsubrutinib 60 mg/upadacitinib placebo -> Elsubrutinib 60 mg/upadacitinib placebo

SUMMARY:
Systemic Lupus Erythematosus (SLE) is an immune-mediated disease associated with inflammation of multiple organ systems. This study will evaluate how well elsubrutinib and upadacitinib given alone or as the ABBV-599 combination (elsubrutinib/upadacitinib) works within the body, in participants who completed study M19-130. This study will assess the change in disease symptoms.

ABBV-599 is an investigational drug being developed for the treatment of Systemic Lupus Erythematosus (SLE). This study is "double-blinded", which means that neither the trial participants nor the study doctors will know who will be given which study drug. Study doctors put the participants into 1 of 4 groups called treatment arms. Each group receives a different treatment. Adult participants with a diagnosis of SLE will be enrolled. Around 260 participants will be enrolled in the study in approximately 100 sites worldwide.

Participants will receive the following for up to 56 weeks:

Participants will receive oral elsubrutinib capsules and/or oral upadacitinib tablets once daily for up to 56 weeks. Participants who were receiving elsubrutinib and/or upadacitnib in M19-130 will continue to receive the same treatment in this study. Participants who were receiving placebo in M19-130 will be re-randomized to one of the 2 combination treatment arms in this study.

Arm 1: Elsubrutinib Dose A and Upadacitinib Dose A Arm 2: Elsubrutinib Dose A and Upadacitinib Dose B

There may be higher burden for participants in this trial compared to their standard of care. Participants will attend monthly visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Completed Study M19-130 (i.e., the randomized controlled trial of elsubrutinib, upadacitinib, and ABBV-599 [elsubrutinib/upadacitinib] combination or matching placebo) and will not have developed any laboratory or clinical discontinuation criteria as defined in that study.
* On stable background treatment for SLE throughout the study.

Exclusion Criteria:

* Active, chronic, or recurrent viral, or bacterial infection.
* Active tuberculosis (TB)
* History of gastrointestinal (GI) perforation, diverticulitis, or a significantly increased risk for GI perforation per investigator assessment.
* Participant require vaccination with live vaccine during study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (87):
- United States (21):
  - Duplicate_AZ Arthritis and Rheumotology Research, PLLC /ID# 227833, Phoenix, Arizona
  - Wallace Rheumatic Studies Center, LLC /ID# 224374, Beverly Hills, California
  - Valerius Medical Group & Research Center /ID# 223922, Los Alamitos, California
  - East Bay Rheumatology Medical /ID# 225493, San Leandro, California
  - University of Colorado Hospital /ID# 245087, Aurora, Colorado
  - Duplicate_Arthritis & Rheumatic Disease Specialties /ID# 227828, Aventura, Florida
  - Millennium Research /ID# 233192, Ormond Beach, Florida
  - IRIS Research and Development, LLC /ID# 227814, Plantation, Florida
  - Deerbrook Medical Associates /ID# 227330, Libertyville, Illinois
  - Qualmedica Research, LLC /ID# 227817, Evansville, Indiana
  - The Center for Rheumatology and Bone Research /ID# 225479, Wheaton, Maryland
  - Beth Israel Deaconess Medical Center /ID# 222505, Boston, Massachusetts
  - June DO, PC /ID# 221841, Lansing, Michigan
  - Duplicate_NYU Langone Health/NYU School of Medicine /ID# 245088, New York, New York
  - STAT Research, Inc. /ID# 221840, Vandalia, Ohio
  - Allegheny Health Network Research Institute /ID# 245086, Pittsburgh, Pennsylvania
  - Dr. Ramesh Gupta /ID# 225524, Memphis, Tennessee
  - Tekton Research, Inc. /ID# 224411, Austin, Texas
  - Accurate Clinical Management /ID# 225509, Houston, Texas
  - SW Rheumatology Res. LLC /ID# 225485, Mesquite, Texas
  - Carilion Clinic /ID# 227832, Roanoke, Virginia
- Argentina (7):
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich /ID# 222569, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Hospital Interzonal General de Agudos General Jose de San Martin /ID# 221893, La Plata, Buenos Aires
  - CER Instituto Medico /ID# 223175, Quilmes, Buenos Aires
  - Aprillus Asistencia e Investigacion /ID# 221890, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto CAICI S.R.L /ID# 221892, Rosario, Santa Fe Province
  - Centro de Investigaciones Medicas Tucuman /ID# 221888, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Clinicas Tucuman /ID# 221889, San Miguel de Tucumán, Tucumán Province
- Australia (3):
  - Rheumatology Research Unit Sunshine Coast /ID# 221816, Maroochydore, Queensland
  - Emeritus Research /ID# 223027, Camberwell, Victoria
  - Monash Medical Centre /ID# 221814, Clayton, Victoria
- Bulgaria (2):
  - UMHAT Sveti Ivan Rilski /ID# 223358, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 223359, Sofia
- China (4):
  - Duplicate_Peking Union Medical College Hospital /ID# 222950, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital /ID# 222851, Guangzhou, Guangdong
  - People's Hospital of Xinjiang /ID# 222928, Urumqi, Guizhou
  - Huashan Hospital, Fudan University /ID# 222929, Shanghai, Shanghai Municipality
- Colombia (5):
  - Duplicate_Centro Integral de Reumatologia del Caribe Circaribe SAS /ID# 221879, Barranquilla, Atlántico
  - Duplicate_Centro de Investigacion en Reumatologia y Especialidades Medicas- CIRE /ID# 221884, Bogota, Cundinamarca
  - Preventive Care Sas /Id# 221881, Chía, Cundinamarca
  - Healthy Medical Center S.A.S /ID# 221882, Zipaquirá, Cundinamarca
  - Clinica Universitaria Bolivari /ID# 221880, Medellin, Valle del Cauca Department
- Germany (2):
  - Duplicate_Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 222963, Berlin
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 222964, Dresden
- Hungary (2):
  - Duplicate_Debreceni Egyetem Klinikai Kozpont /ID# 222480, Debrecen, Hajdú-Bihar
  - Vital Medicina Kft /ID# 222479, Veszprém, Veszprém megye
- Duplicate_Azienda Ospedaliero-Universitaria di Ferrara-Arcispedale Sant Anna /ID# 221919, Cona, Ferrara, Italy
- Japan (10):
  - Chukyo Hospital /ID# 223398, Nagoya, Aichi-ken
  - NHO Nagoya Medical Center /ID# 222397, Nagoya, Aichi-ken
  - Hospital of the University of Occupational and Environmental Health, Japan /ID# 222499, Kitakyushu-shi, Fukuoka
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital /ID# 222393, Hiroshima, Hiroshima
  - National Hospital Organization Asahikawa Medical Center /ID# 222394, Asahikawa-shi, Hokkaido
  - EIRAKU Internal Medicine Clinic /ID# 222385, Kagoshima, Kagoshima-ken
  - Tohoku University Hospital /ID# 222392, Sendai, Miyagi
  - Shinshu University Hospital /ID# 222395, Matsumoto-shi, Nagano
  - Saitama Medical Center /ID# 222389, Kawagoe-shi, Saitama
  - Keio University Hospital /ID# 222498, Shinjuku-ku, Tokyo
- Mexico (6):
  - Morales Vargas Centro de Investigacion S.C. /ID# 221912, León, Guanajuato
  - Centro Integral en Reumatologia S.A de C.V /ID# 221914, Guadalajara, Jalisco
  - Centro de Estudios de Investigación Básica y Clínica, S.C. /ID# 221910, Guadalajara, Jalisco
  - RM Pharma Specialists S.A de C.V. /ID# 221915, Mexico City, Mexico City
  - CINTRE, Centro de Investigación y Tratamiento Reumatológico SC /ID# 221913, Mexico City, Mexico City
  - Medical Care & Research SA de CV /ID# 221911, Mérida, Yucatán
- North Shore Hospital /ID# 221850, Takapuna, Auckland, New Zealand
- Poland (4):
  - Ortopedyczno-Rehabilitacyjny Szpital Kliniczny im. Wiktora Degi /ID# 221859, Poznan, Greater Poland Voivodeship
  - Centrum Nowoczesnych Terapii Dobry Lekarz Sp. z o.o. /ID# 224430, Krakow, Lesser Poland Voivodeship
  - WroMedica I. Bielicka, A. Strzalkowska s.c. /ID# 221860, Wroclaw, Lower Silesian Voivodeship
  - MTZ Clinical Research Powered by Pratia /ID# 224431, Warsaw, Masovian Voivodeship
- Puerto Rico (2):
  - GCM Medical Group PSC /ID# 224394, San Juan
  - Mindful Medical Research /ID# 222513, San Juan
- Seoul National University Hospital /ID# 221897, Seoul, Seoul Teugbyeolsi, South Korea
- Spain (8):
  - HUA - Txagorritxu /ID# 221992, Vitoria-Gasteiz, Alava
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 221995, Sabadell, Barcelona
  - Hospital Universitario Basurto /ID# 221999, Bilbao, Vizcaya
  - Hospital Universitario de Galdakao /ID# 221996, Galdakao, Vizcaya
  - Duplicate_Hospital Universitario A Coruna - CHUAC /ID# 221993, A Coruña
  - Hospital Universitario 12 de Octubre /ID# 221994, Madrid
  - Hospital Universitario Virgen de Valme /ID# 221997, Seville
  - Hospital Universitario y Politecnico La Fe /ID# 221998, Valencia
- Taiwan (6):
  - Taichung Veterans General Hospital /ID# 221748, Taichung, Keelung
  - Taipei Veterans General Hosp /ID# 221746, Taipei, Keelung
  - National Taiwan University Hospital /ID# 221745, Taipei City, Taipei
  - China Medical University Hospital /ID# 221747, Taichung
  - Taipei Medical University Hospital /ID# 227653, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 222469, Taoyuan
- United Kingdom (2):
  - Guys and St Thomas NHS Foundation Trust /ID# 221863, London, London, City of
  - Duplicate_Manchester University NHS Foundation Trust /ID# 221861, Manchester

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set (FAS): all participants who received at least 1 dose of study drug in Study M20-186. Participants are grouped according to treatment sequence as randomized for Studies M19-130 and M20-186.
Period: Overall Study
Arm/Group | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) -> ABBV-599 High Dose | Elsubrutinib Placebo/Upadacitinib 30 mg -> Elsubrutinib Placebo/Upadacitinib 30 mg | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 High Dose | ABBV-599 Low Dose (Elsubrutinib 60 mg/Upadacitinib 15 mg) -> ABBV-599 Low Dose | Elsubrutinib 60 mg/Upadacitinib Placebo -> Elsubrutinib 60 mg/Upadacitinib Placebo | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 Low Dose
Started | 45 | 47 | 35 | 19 | 25 | 14
Completed | 41 | 38 | 31 | 6 | 1 | 1
Not Completed | 4 | 9 | 4 | 13 | 24 | 13
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 2 | 7 | 2 | 1 | 1 | 0
Not completed — Other, not specified | 1 | 2 | 1 | 0 | 0 | 1
Not completed — Sponsor decision based on interim analysis data review | 0 | 0 | 0 | 11 | 23 | 9

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants who received at least 1 dose of study drug in Study M20-186. Participants are grouped according to treatment sequence as randomized for Studies M19-130 and M20-186. Per protocol, demographic and baseline characteristics are summarized as measured at the start of Study M19-130.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) -> ABBV-599 High Dose | Elsubrutinib Placebo/Upadacitinib 30 mg -> Elsubrutinib Placebo/Upadacitinib 30 mg | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 High Dose | ABBV-599 Low Dose (Elsubrutinib 60 mg/Upadacitinib 15 mg) -> ABBV-599 Low Dose | Elsubrutinib 60 mg/Upadacitinib Placebo -> Elsubrutinib 60 mg/Upadacitinib Placebo | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 Low Dose | Total
Number analyzed (Participants) | 45 | 47 | 35 | 19 | 25 | 14 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (11.39) | 42.5 (12.00) | 40.6 (11.75) | 38.3 (10.52) | 41.2 (11.60) | 42.5 (11.57) | 41.6 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 35 | 18 | 24 | 14 | 175
  Male | 3 | 5 | 0 | 1 | 1 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 2 | 1 | 2 | 0 | 8
  Asian | 6 | 10 | 12 | 6 | 3 | 2 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 6 | 0 | 1 | 1 | 1 | 11
  White | 32 | 26 | 20 | 10 | 16 | 10 | 114
  More than one race | 2 | 5 | 1 | 1 | 3 | 1 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs) are defined as an adverse event with an onset date that is on or after the first dose of study drug from Study M20-186, and no more than 30 days after the last dose of study drug from Study M20-186. For more details on adverse events please see the Adverse Event section.
Time Frame: From the first dose of study drug in Study M20-186 up to 30 days after the last dose of study drug, up to 442 days
Population: Safety analysis set: all participants who received at least 1 dose of study drug in Study M20-186, grouped according to treatment sequence actually received
Measure: Number; unit: participants
Arm/Group | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) -> ABBV-599 High Dose | Elsubrutinib Placebo/Upadacitinib 30 mg -> Elsubrutinib Placebo/Upadacitinib 30 mg | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 High Dose | ABBV-599 Low Dose (Elsubrutinib 60 mg/Upadacitinib 15 mg) -> ABBV-599 Low Dose | Elsubrutinib 60 mg/Upadacitinib Placebo -> Elsubrutinib 60 mg/Upadacitinib Placebo | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 Low Dose
Number analyzed (Participants) | 45 | 47 | 35 | 19 | 25 | 14
participants
  Any TEAE | 34 | 31 | 30 | 11 | 11 | 7
  TESAE | 5 | 5 | 1 | 2 | 1 | 2

2. Secondary Outcome: Percentage of Participants Achieving Systemic Lupus Erythematosus (SLE) Responder Index (SRI)-4
Description: SLE Responder Index (SRI)-4 is defined as follows with all criteria compared to Baseline in Study M19-130:
  * ≥4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score
  * No worsening of the overall condition (< 0.3 point increase in Physician's Global Assessment [PhGA])
  * No new British Isles Lupus Assessment Group (BILAG) A or more than 1 new BILAG B disease activity scores (i.e., no organ system changes from baseline B/C/D/E to A and no more than 1 organ system changes from baseline C/D/E to B). A letter score is assigned to each organ system with following indications: A = severe, B = moderate, C = mild, D = inactive with prior history, and E = inactive with no history.
Time Frame: Baseline of Study M19-130 (Week 0), Weeks 56, 64, 72, 80, 88, 96, 104
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug in Study M20-186; as observed (AO) analysis. When 50% of planned participants in Study M19-130 had completed Week 24 or withdrawn from the study, the ABBV-599 Low Dose and elsubrutinib 60 mg treatment groups were terminated as these groups did not meet projected efficacy. Per protocol, terminated groups were removed from the efficacy analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) -> ABBV-599 High Dose | Elsubrutinib Placebo/Upadacitinib 30 mg -> Elsubrutinib Placebo/Upadacitinib 30 mg | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 High Dose
Number analyzed (Participants) | 45 | 46 | 35
percentage of participants
  Week 56 | 71.1 [57.9 to 84.4] | 76.1 [63.8 to 88.4] | 54.3 [37.8 to 70.8]
  Week 64: number analyzed (Participants) | 44 | 45 | 34
  Week 64 | 70.5 [57.0 to 83.9] | 75.6 [63.0 to 88.1] | 58.8 [42.3 to 75.4]
  Week 72: number analyzed (Participants) | 41 | 45 | 34
  Week 72 | 80.5 [68.4 to 92.6] | 88.9 [79.7 to 98.1] | 64.7 [48.6 to 80.8]
  Week 80: number analyzed (Participants) | 40 | 45 | 33
  Week 80 | 75.0 [61.6 to 88.4] | 82.2 [71.1 to 93.4] | 57.6 [40.7 to 74.4]
  Week 88: number analyzed (Participants) | 40 | 42 | 33
  Week 88 | 82.5 [70.7 to 94.3] | 85.7 [75.1 to 96.3] | 48.5 [31.4 to 65.5]
  Week 96: number analyzed (Participants) | 41 | 39 | 32
  Week 96 | 82.9 [71.4 to 94.4] | 76.9 [63.7 to 90.1] | 62.5 [45.7 to 79.3]
  Week 104: number analyzed (Participants) | 41 | 39 | 31
  Week 104 | 85.4 [74.5 to 96.2] | 82.1 [70.0 to 94.1] | 61.3 [44.1 to 78.4]

3. Secondary Outcome: Percentage of Participants Achieving British Isles Lupus Assessment Group (BILAG)-Based Combined Lupus Assessment (BICLA) Response
Description: BICLA is a composite responder index. Achievement of BICLA response is defined as improvement in all initial A and B BILAG scores, with no more than one new BILAG B score without worsening of the overall condition (no worsening in Physician's Global Assessment [PhGA], < 0.3 point increase) and no worsening of the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score.
Time Frame: Baseline of Study M19-130 (Week 0), Weeks 56, 64, 72, 80, 88, 96, 104
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) -> ABBV-599 High Dose | Elsubrutinib Placebo/Upadacitinib 30 mg -> Elsubrutinib Placebo/Upadacitinib 30 mg | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 High Dose
Number analyzed (Participants) | 45 | 46 | 35
percentage of participants
  Week 56 | 73.3 [60.4 to 86.3] | 67.4 [53.8 to 80.9] | 60.0 [43.8 to 76.2]
  Week 64: number analyzed (Participants) | 44 | 45 | 34
  Week 64 | 75.0 [62.2 to 87.8] | 84.4 [73.9 to 95.0] | 55.9 [39.2 to 72.6]
  Week 72: number analyzed (Participants) | 41 | 45 | 34
  Week 72 | 73.2 [59.6 to 86.7] | 88.9 [79.7 to 98.1] | 61.8 [45.4 to 78.1]
  Week 80: number analyzed (Participants) | 40 | 45 | 33
  Week 80 | 70.0 [55.8 to 84.2] | 77.8 [65.6 to 89.9] | 57.6 [40.7 to 74.4]
  Week 88: number analyzed (Participants) | 40 | 42 | 33
  Week 88 | 80.0 [67.6 to 92.4] | 85.7 [75.1 to 96.3] | 57.6 [40.7 to 74.4]
  Week 96: number analyzed (Participants) | 41 | 39 | 32
  Week 96 | 78.0 [65.4 to 90.7] | 76.9 [63.7 to 90.1] | 59.4 [42.4 to 76.4]
  Week 104: number analyzed (Participants) | 41 | 39 | 31
  Week 104 | 78.0 [65.4 to 90.7] | 69.2 [54.7 to 83.7] | 54.8 [37.3 to 72.4]

4. Secondary Outcome: Change From Baseline in Daily Prednisone Dose Over Time
Description: Participants'current use of steroid therapy was assessed at each study visit, and the amount of daily prednisone was documented.
Time Frame: Baseline of M19-130 (Week 0), Weeks 56, 64, 72, 80, 88, 96, 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) -> ABBV-599 High Dose | Elsubrutinib Placebo/Upadacitinib 30 mg -> Elsubrutinib Placebo/Upadacitinib 30 mg | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 High Dose
Number analyzed (Participants) | 45 | 47 | 35
mg
  Week 56 | -3.9 (5.96) | -3.5 (5.99) | -4.9 (6.99)
  Week 64: number analyzed (Participants) | 45 | 46 | 35
  Week 64 | -4.2 (5.51) | -3.7 (5.97) | -5.0 (6.87)
  Week 72: number analyzed (Participants) | 42 | 46 | 34
  Week 72 | -4.0 (6.59) | -4.9 (7.23) | -5.2 (6.88)
  Week 80: number analyzed (Participants) | 41 | 45 | 34
  Week 80 | -5.1 (5.96) | -4.4 (8.05) | -5.2 (6.88)
  Week 88: number analyzed (Participants) | 41 | 42 | 33
  Week 88 | -5.5 (5.83) | -5.2 (6.02) | -6.2 (7.04)
  Week 96: number analyzed (Participants) | 41 | 40 | 32
  Week 96 | -5.5 (5.88) | -5.7 (5.78) | -7.3 (6.54)
  Week 104: number analyzed (Participants) | 41 | 39 | 31
  Week 104 | -5.8 (6.02) | -5.5 (5.65) | -7.7 (6.64)

5. Secondary Outcome: Number of Flares Per Patient-year by Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA) SLE Disease Activity Index (SLEDAI) Flare Index Through Week 104
Description: The SELENA SLEDAI flare index defines mild/moderate or severe SLE flares using the SLEDAI score, definitions of worsening signs and symptoms, treatment changes, and Physician's Global Assessment of Disease Activity.
Time Frame: From Week 56 through Week 104
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events per patient-year
Arm/Group | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) -> ABBV-599 High Dose | Elsubrutinib Placebo/Upadacitinib 30 mg -> Elsubrutinib Placebo/Upadacitinib 30 mg | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 High Dose
Number analyzed (Participants) | 45 | 47 | 35
Events per patient-year
  Mild/Moderate | 0.62 [0.39 to 0.84] | 1.41 [1.06 to 1.75] | 1.39 [0.99 to 1.78]
  Severe | 0.00 [0.00 to 0.00] | 0.04 [-0.02 to 0.10] | 0.17 [0.03 to 0.31]
  Overall | 0.62 [0.39 to 0.84] | 1.45 [1.10 to 1.80] | 1.56 [1.14 to 1.97]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events were collected from the time informed consent was signed through the end of the study. Median time on follow-up was for 422 days for the ABBV-599 High -> ABBV-599 High group; 423 days for the Upa -> Upa and Pbo -> ABBV-599 High groups; 245 days for the ABBV-599 Low -> ABBV-599 Low group; 163 days for the Els -> Els group; and 142.5 days for the Pbo -> ABBV-599 Low group.
Arm/Group | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) -> ABBV-599 High Dose | Elsubrutinib Placebo/Upadacitinib 30 mg -> Elsubrutinib Placebo/Upadacitinib 30 mg | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 High Dose | ABBV-599 Low Dose (Elsubrutinib 60 mg/Upadacitinib 15 mg) -> ABBV-599 Low Dose | Elsubrutinib 60 mg/Upadacitinib Placebo -> Elsubrutinib 60 mg/Upadacitinib Placebo | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 Low Dose
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/47 | 0/35 | 0/19 | 0/25 | 0/14
Serious Adverse Events (participants affected / at risk) | 5/45 | 5/47 | 1/35 | 2/19 | 1/25 | 2/14
Other Adverse Events (participants affected / at risk) | 24/45 | 18/47 | 30/35 | 11/19 | 4/25 | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) -> ABBV-599 High Dose (N=45) | Elsubrutinib Placebo/Upadacitinib 30 mg -> Elsubrutinib Placebo/Upadacitinib 30 mg (N=47) | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 High Dose (N=35) | ABBV-599 Low Dose (Elsubrutinib 60 mg/Upadacitinib 15 mg) -> ABBV-599 Low Dose (N=19) | Elsubrutinib 60 mg/Upadacitinib Placebo -> Elsubrutinib 60 mg/Upadacitinib Placebo (N=25) | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 Low Dose (N=14)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEROSITIS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKULL FRACTURED BASE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL HAEMATOMA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) -> ABBV-599 High Dose (N=45) | Elsubrutinib Placebo/Upadacitinib 30 mg -> Elsubrutinib Placebo/Upadacitinib 30 mg (N=47) | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 High Dose (N=35) | ABBV-599 Low Dose (Elsubrutinib 60 mg/Upadacitinib 15 mg) -> ABBV-599 Low Dose (N=19) | Elsubrutinib 60 mg/Upadacitinib Placebo -> Elsubrutinib 60 mg/Upadacitinib Placebo (N=25) | Elsubrutinib Placebo/Upadacitinib Placebo -> ABBV-599 Low Dose (N=14)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TYPE V HYPERLIPIDAEMIA (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GRANULOMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 11 (11) | 7 (7) | 0 (0) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
MYCOPLASMA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TINEA PEDIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
TINEA VERSICOLOUR (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (5) | 3 (4) | 6 (7) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 7 (9) | 3 (7) | 6 (8) | 3 (4) | 1 (1) | 1 (1)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
IMMUNISATION REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
LUPUS NEPHRITIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUS PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CUTANEOUS VASCULITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT04451772/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT04451772/SAP_001.pdf